CLINICAL TRIAL: NCT02993536
Title: Clonal Evolution of B Cells in High-risk Chronic Lymphocytic Leukemia Patients After Idelalisib-rituximab Treatment
Brief Title: Clonal Evolution of B Cells in High-risk CLL After Idelalisib-rituximab
Status: Withdrawn | Type: Observational
Why Stopped: Low likelihood to usedrug in clinic practice based on emergining AE profile and data from front line clinical trials
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 30415
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Biospecimen Collection

SUMMARY:
The purpose of the study is to assess the evolution of B cells at a genetic and surface-marker level in high-risk CLL after idelalisib-rituximab treatment. The targeted population includes 20 subjects ages 18 or older diagnosed with high-risk CLL. This will include patients with relapsed or refractory disease who require therapy with idelalisib and rituximab as per FDA label. This is an observational study for peripheral blood samples of these patients collected at pre-determined time points.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Ability to provide informed consent
* Ability to provide peripheral blood samples
* Diagnosis of CLL
* Indication(s) for CLL therapy
* At least one criterion for high-risk disease

  * Disease refractory (e.g., no response) to at least one round of chemotherapy
  * Disease that has relapsed (i.e., returned) after at least one round of chemotherapy
  * Proven presence of the 17p deletion within CLL cells
* Planned receipt of idelalisib-rituximab as per FDA guidelines and patient's oncologists

Exclusion Criteria:

* Patients who do not meet the diagnostic criteria for CLL or at least one indication for treatment.
* Patients who are receiving idelalisib with an off-label indication
* Patients who do not or cannot provide informed consent to donate peripheral blood tumor samples to our stem cell core facility
* Patients who do not provide informed consent to collect clinical, prognostic, and outcomes data during the time period that they are treated with idelalisib-rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with relapsed or refractory CLL requiring treatment and receiving idelalisib-rituximab
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Estimated); Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Number of somatic hypermutation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mato, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States